CLINICAL TRIAL: NCT04311671
Title: A Randomized, Double Blind, Parallel Group Clinical Trial to Evaluate the Safety of Moxidectin Compared With Ivermectin in Individuals Living in Onchocerciasis Endemic Areas and in Individuals Living in Onchocerciasis Endemic Areas With High Levels of Lymphatic Filariasis Co-endemicity Receiving Concomitant Treatment With Albendazole
Brief Title: Safety of a Single Dose of Moxidectin Compared With Ivermectin in Individuals Living in Onchocerciasis Endemic Areas and in Individuals Living in Onchocerciasis Endemic Areas With High Levels of Lymphatic Filariasis Co-endemicity Receiving Concomitant Albendazole
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medicines Development for Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDGH-MOX-3002
Record Dates: First submitted 2020-03-14; First posted 2020-03-17 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Onchocerciasis
MeSH Terms: conditions — Onchocerciasis | interventions — moxidectin; Ivermectin; Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Moxidectin (Experimental): In onchocerciasis endemic areas: Moxidectin 8 mg per oral on Day 0
  Interventions: Drug: Moxidectin
- Ivermectin (Active Comparator): In onchocerciasis endemic areas: Ivermectin treatment with approximately 150 µg/kg per oral determined based on height on Day 0
  Interventions: Drug: Ivermectin
- Moxidectin with concomitant Albendazole (Experimental): In onchocerciasis endemic areas with high levels of lymphatic filariasis co-endemicity: Moxidectin 8 mg per oral with concomitant albendazole 400 mg per oral on Day 0
  Interventions: Drug: Moxidectin; Drug: Albendazole
- Ivermectin with concomitant Albendazole (Active Comparator): In onchocerciasis endemic areas with high levels of lymphatic filariasis co-endemicity: Ivermectin treatment with approximately 150 microgram/kilogram (μg/kg) per oral determined based on height with concomitant albendazole 400 mg per oral on Day 0
  Interventions: Drug: Ivermectin; Drug: Albendazole

INTERVENTIONS:
Drug: Moxidectin — 2 mg tablets, encapsulated for blinding
  Arms: Moxidectin; Moxidectin with concomitant Albendazole
Drug: Ivermectin — 3 mg tablets, encapsulated for blinding
  Arms: Ivermectin; Ivermectin with concomitant Albendazole
Drug: Albendazole — 400 mg tablets
  Arms: Ivermectin with concomitant Albendazole; Moxidectin with concomitant Albendazole

SUMMARY:
The purpose of this phase 3b study is to determine the safety of a single dose of moxidectin, compared to a single dose of ivermectin, in individuals living in onchocerciasis endemic areas and in individuals living in onchocerciasis endemic areas with high levels of lymphatic filariasis co-endemicity receiving concomitant albendazole.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent, or assent with parental or guardian written consent*
2. Known O. volvulus skin microfilariae density ≥0 microfilariae/mg skin (participants ≥12 years of age only).
3. Living in an onchocerciasis endemic area.
4. Age ≥4 years
5. All female participants of childbearing potential must commit to the use of a reliable method of birth control until 3 months after administration of investigational product (Month 3). * Expression of 'deliberate objection' will be the basis for assessing assent of children aged ≥ 4 to <6 years

Exclusion Criteria:

1. Pregnant or breast-feeding.
2. Any concurrent condition that, in the opinion of the Investigator, would preclude evaluation of response to treatment or would pose undue risk to the participant's health.
3. Has received ivermectin or oral diethylcarbamazine (DEC) within 30 days of Baseline.
4. Has received treatment with an investigational agent within the 30 days (or 5 half-lives, whichever is longer) prior to planned investigational product administration.
5. Known or suspected allergy to ivermectin or moxidectin or their excipients and, in areas with high levels of LF co-endemicity, known or suspected allergy to albendazole and its excipients.
6. Self-reported planned or ongoing activities within the study period that would make it unlikely that the participant will be available for follow-up examinations.
7. Infection with Loa loa.
8. Height <90 cm.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12979 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Ukety, MD, DO, MPH, Principal Investigator — Centre de Recherche en Maladies Tropicales de l'Ituri; Benjamin Koudou, PhD, Principal Investigator — Centre Suisse de Recherches Scientifiques en Coˆte d'Ivoire
Locations (2):
- Centre Suisse de Recherches Scientifiques en Coˆte d'Ivoire, Abidjan, Côte d’Ivoire
- Centre de Recherche pour les Maladies Tropicales Negligees, Rethy, Ituri, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Moxidectin: Participants randomized in a blinded fashion to this group received treatment with a single oral dose of moxidectin as 4 x 2mg tablet-in-capsules for adults and children from 8 years. Children < 12 years received the required number of tablets removed from the capsules and without placebo, administered by an unblinded pharmacist or staff member not involved in the outcomes assessment of participants. Children aged 4 to less than 8 years received treatment with 2 x 2mg moxidectin tablets.
- Ivermectin: Participants randomized in a blinded fashion to this group received treatment with a single dose of ivermectin of approximately 150mcg/kg, estimated by height, administered as 3mg ivermectin tablet-in-capsules plus placebo to match (total 4 capsules): Height 90-119cm (1 x 3mg); 120 to 139cm (2 x 3mg); 140 to 159cm (3 x 3mg); > 159cm (4 x 3mg) tablets in capsules. Children < 12 years received the required number of tablets removed from the capsules and without placebo, administered by an unblinded pharmacist or staff member not involved in assessment of participants.
- Moxidectin Plus Albendazole: Participants randomized in a blinded fashion to this group received treatment with a single oral dose of moxidectin as 4 x 2mg tablet-in-capsules for adults and children from 8 years. Children < 12 years received the required number of tablets removed from the capsules and without placebo, administered by an unblinded pharmacist or staff member not involved in the outcomes assessment of participants. Children aged 4 to less than 8 years received treatment with 2 x 2mg moxidectin tablets. All participants received a single Albendazole tablet 400mg as a single open label dose concurrently with moxidectin.
- Ivermectin Plus Albendazole: Participants randomized in a blinded fashion to this group received treatment with a single oral dose of moxidectin as 4 x 2mg tablet-in-capsules for adults and children from 8 years. Children < 12 years received the required number of tablets removed from the capsules and without placebo, administered by an unblinded pharmacist or staff member not involved in the outcomes assessment of participants. Children aged 4 to less than 8 years received treatment with 2 x 2mg moxidectin tablets. All participants received a single Albendazole tablet 400mg as a single open label dose concurrently with ivermectin.
Period: Overall Study
Arm/Group | Moxidectin | Ivermectin | Moxidectin Plus Albendazole | Ivermectin Plus Albendazole
Started | 6421 (Treated population) | 1605 (Treated population) | 3959 (Treated population) | 994 (Treated population)
Completed | 6395 | 1592 | 3891 | 977
Not Completed | 26 | 13 | 68 | 17

BASELINE CHARACTERISTICS:
Groups:
- Moxidectin: In onchocerciasis endemic areas: Moxidectin 8 mg per oral on Day 0 for adults and children from 8 years, 4 mg for children 4 to < 8 years.
  Moxidectin: 2 mg tablets, encapsulated for blinding
- Moxidectin With Concomitant Albendazole: In onchocerciasis endemic areas with high levels of lymphatic filariasis co-endemicity: Moxidectin 8 mg per oral for adults and children from 8 years, 4 mg for children 4 to < 8 years, with concomitant albendazole 400 mg per oral on Day 0
  Moxidectin: 2 mg tablets, encapsulated for blinding
  Albendazole: 400 mg tablets
- Total: Total of all reporting groups
Arm/Group | Moxidectin | Ivermectin | Moxidectin With Concomitant Albendazole | Ivermectin With Concomitant Albendazole | Total
Number analyzed (Participants) | 6421 | 1605 | 3959 | 994 | 12979
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2015 | 461 | 1387 | 340 | 4203
  Between 18 and 65 years | 4069 | 1061 | 2409 | 610 | 8149
  >=65 years | 337 | 83 | 163 | 44 | 627
Age, Continuous [Mean (Full Range); unit: years] | 30.4 [4 to 93] | 31.2 [4 to 84] | 28.5 [4 to 91] | 28.6 [4 to 96] | 29.8 [4 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2954 | 724 | 1829 | 470 | 5977
  Male | 3467 | 881 | 2130 | 524 | 7002
Race/Ethnicity, Customized [Number; unit: participants] — All participants were recruited from villages in rural areas of the Democratic Republic of Congo (Ituri province) and from the Akoupe region in Cote D'Ivoire. Only people of black African race were enrolled.
  participants
    Race - Black African | 6421 | 1605 | 3959 | 994 | 12979
Region of Enrollment [Number; unit: participants]
  Congo, The Democratic Republic of the | 6421 | 1605 | 0 | 0 | 8026
  Côte D'Ivoire | 0 | 0 | 3959 | 994 | 4953
Number of Participants with Onchocerca volvulus skin microfilariae (mf) [Number; unit: participants] — Assessment for presence of O. volvulus skin microfilariae in participants 12 years and older. Two (2) skin snips, one taken from each iliac crest, were collected prior to treatment by corneoscleral punch, processed in saline and the emerging microfilariae counted (if present). The results were then standardized to the number of microfilariae per milligram of skin Population: Only participants 12 years and older had skin microfilariae (mf) measured, hence the total number of participants assessed as having undetectable or detectable skin mf (n=11947) is less than the overall study population (n=12979), a difference of 1032 (children under 12 years)
  participants
    Overall tested: number analyzed (Participants) | 6271 | 1568 | 3282 | 826 | 11947
    Overall tested | 6271 | 1568 | 3282 | 826 | 11947
    Undetectable (skin mf =0): number analyzed (Participants) | 6271 | 1568 | 3282 | 826 | 11947
    Undetectable (skin mf =0) | 6065 | 1509 | 3067 | 751 | 11392
    Detectable (skin mf>0): number analyzed (Participants) | 6271 | 1568 | 3282 | 826 | 11947
    Detectable (skin mf>0) | 206 | 59 | 215 | 75 | 555
Number of participants with LF antigenemia and/or microfilaremia [Number; unit: participants] — Assessment for presence of circulating lymphatic filarial antigen (CFA) was conducted using a semiquantitative rapid filarial test strip. A nocturnal venous blood sample was then collected for assessment of microfilaremia in participants with a CFA result greater than 0. This test was only conducted in the Cote D'Ivoire region where LF was was known to be endemic. Population: This assessment was only conducted in the Cote D'Ivoire region where LF was was known to be endemicand only in participants aged 12 years and older. Hence only participants in the Moxidectin plus Albendazole or the Ivermectin plus Albendazole arms have results for this measure
  participants
    CFA Positive (Category 1-3) with or without microfilaremia: number analyzed (Participants) | 0 | 0 | 3286 | 826 | 4112
    CFA Positive (Category 1-3) with or without microfilaremia |  |  | 107 | 23 | 130
    CFA negative: number analyzed (Participants) | 0 | 0 | 3286 | 826 | 4112
    CFA negative |  |  | 3179 | 803 | 3982

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Treatment Emergent Adverse Events
Description: Participant incidence rates of treatment emergent adverse events following a single dose of moxidectin versus a single dose of ivermectin will be assessed separately by endemic area. Treatment emergent adverse events may also be pooled across both endemic areas (pooled monotherapy and combination therapies separately for moxidectin and ivermectin), provided a qualitative assessment shows they are similar enough to enable the interpretation of the pooled analysis.
Time Frame: Up to 3 months
Population: Participants who received a single dose of moxidectin or ivermectin and participants who received a single dose of moxidectin or ivermectin with albendazole analyzed separately by endemic area and pooled.
Measure: Number; unit: participants
Groups:
- Moxidectin +/- Albendazole (Pooled): Participants randomized in a blinded fashion to this group received treatment with a single oral dose of moxidectin as 4 x 2mg tablet-in-capsules for adults and children from 8 years. Children < 12 years received the required number of tablets removed from the capsules and without placebo, administered by an unblinded pharmacist or staff member not involved in the outcomes assessment of participants. Children aged 4 to less than 8 years received treatment with 2 x 2mg moxidectin tablets. Participants received treatment with or without a single Albendazole tablet 400mg as a single open label dose concurrently with moxidectin, depending on LF-endemicity in the area
- Ivermectin +/- Albendazole (Pooled): Participants randomized in a blinded fashion to this group received treatment with a single oral dose of moxidectin as 4 x 2mg tablet-in-capsules for adults and children from 8 years. Children < 12 years received the required number of tablets removed from the capsules and without placebo, administered by an unblinded pharmacist or staff member not involved in the outcomes assessment of participants. Children aged 4 to less than 8 years received treatment with 2 x 2mg moxidectin tablets. Participants received treatment with or without a single Albendazole tablet 400mg as a single open label dose concurrently with ivermectin, depending on LF-endemicity in the area
Arm/Group | Moxidectin | Ivermectin | Moxidectin Plus Albendazole | Ivermectin Plus Albendazole | Moxidectin +/- Albendazole (Pooled) | Ivermectin +/- Albendazole (Pooled)
Number analyzed (Participants) | 6421 | 1605 | 3959 | 994 | 10380 | 2599
participants
  Number of Participants with one or more Treatment Emergent Adverse Events (TEAEs) | 346 | 79 | 1199 | 288 | 1545 | 367
  Number of Participants with one or more TEAEs defined as a Mazzotti Reaction | 173 | 47 | 455 | 98 | 628 | 145
  Number of Participants with Severe (Gr 3 or 4) TEAE | 18 | 5 | 66 | 14 | 84 | 19
  Number of Participants with TEAE defined as Serious | 18 | 4 | 4 | 0 | 22 | 4
  Number of participants with TEAE leading to Death | 6 | 2 | 3 | 0 | 9 | 2
  Number of Participants with a TEAE considered Related to Moxidectin or Ivermectin | 189 | 50 | 576 | 128 | 765 | 178
  Number of Participants with a Severe TEAE considered Related to Moxidectin or Ivermectin | 0 | 0 | 0 | 0 | 0 | 0
  Number of Participants with a TEAE considered Related to Albendazole | 0 | 0 | 34 | 7 | 34 | 7
  Number of Participants with a Severe TEAE considered Related to Albendazole | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all participants daily for 5 days and up to 3 months after treatment. More than 98% of participants completed a Month 3 visit.
Description: Adverse events were recorded by the Investigator and may have been initially recorded at a local health center a participant choose to attend or by a study team member during the protocol scheduled follow up visits or ad hoc visits at the request of a participant.
Arm/Group | Moxidectin | Ivermectin | Moxidectin Plus Albendazole | Ivermectin Plus Albendazole | Moxidectin +/- Albendazole (Pooled) | Ivermectin +/- Albendazole (Pooled)
All-Cause Mortality (participants affected / at risk) | 6/6421 | 2/1605 | 3/3959 | 0/994 | 9/10380 | 2/2599
Serious Adverse Events (participants affected / at risk) | 18/6421 | 4/1605 | 4/3959 | 0/994 | 22/10380 | 4/2599
Other Adverse Events (participants affected / at risk) | 346/6421 | 79/1605 | 1199/3959 | 288/994 | 1545/10380 | 367/2599
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxidectin (N=6421) | Ivermectin (N=1605) | Moxidectin Plus Albendazole (N=3959) | Ivermectin Plus Albendazole (N=994) | Moxidectin +/- Albendazole (Pooled) (N=10380) | Ivermectin +/- Albendazole (Pooled) (N=2599)
Cardiac Failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polydactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastritis hemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complicated malaria or malaria (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Giardiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fournier's gangrene (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxidectin (N=6421) | Ivermectin (N=1605) | Moxidectin Plus Albendazole (N=3959) | Ivermectin Plus Albendazole (N=994) | Moxidectin +/- Albendazole (Pooled) (N=10380) | Ivermectin +/- Albendazole (Pooled) (N=2599)
Tachycardia or Palpitations (Cardiac disorders) | 5 (5) | 1 (1) | 7 (7) | 2 (2) | 12 (12) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 6 (6) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 6 (6) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 10 (10) | 0 (0) | 12 (12) | 0 (0)
Conjunctival/ocular hyperemia or conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 14 (14) | 1 (1) | 14 (14) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 9 (9) | 2 (2) | 10 (10) | 2 (2)
Eye pruritis (Eye disorders) | 0 (0) | 0 (0) | 25 (27) | 7 (8) | 25 (27) | 7 (8)
Lacrimation increased (Eye disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 2 (2)
Abdominal pain and/or distension (Gastrointestinal disorders) | 11 (11) | 0 (0) | 62 (62) | 20 (20) | 73 (73) | 20 (20)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 2 (2) | 57 (60) | 16 (16) | 64 (67) | 18 (18)
Constipation / Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 8 (8) | 1 (1) | 8 (8) | 1 (1)
Gastritis (Gastrointestinal disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Nausea and/or vomiting (Gastrointestinal disorders) | 6 (6) | 2 (2) | 10 (10) | 1 (1) | 12 (12) | 3 (3)
Fatigue or Asthenia (General disorders) | 5 (5) | 4 (4) | 21 (22) | 5 (5) | 26 (27) | 9 (9)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 0 (0)
Influenza-like illness, chills or pyrexia (General disorders) | 2 (2) | 0 (0) | 38 (38) | 8 (8) | 40 (40) | 8 (8)
Chest pain (General disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 6 (6) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 28 (28) | 3 (3) | 28 (28) | 3 (3)
Peripheral swelling / swelling (General disorders) | 0 (0) | 0 (0) | 33 (34) | 9 (9) | 33 (34) | 9 (9)
Malaria / complicated malaria (Infections and infestations) | 50 (51) | 9 (10) | 232 (243) | 66 (71) | 282 (294) | 75 (81)
Infections (various, not malaria) (Infections and infestations) | 24 (24) | 4 (4) | 89 (98) | 16 (16) | 113 (122) | 20 (20)
Injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 22 (23) | 7 (8) | 23 (24) | 8 (9) — Abrasions, snake bite, wounds, joint injuries
Appetite - disorder / decreased (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 3 (3) — One case of hyperphagia (MOX+ALB)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0) | 17 (17) | 5 (5) | 24 (24) | 5 (5)
Back or neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 33 (34) | 6 (6) | 37 (38) | 8 (8)
Joint swelling / limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (5) | 3 (3) | 2 (5)
Myalgia / musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 9 (9) | 2 (2) | 39 (39) | 7 (7) | 48 (48) | 9 (9)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 12 (12) | 3 (4) | 13 (13) | 3 (4)
Dizziness (Nervous system disorders) | 6 (6) | 4 (4) | 11 (11) | 3 (3) | 17 (17) | 7 (7)
Headache (Nervous system disorders) | 84 (84) | 21 (21) | 161 (168) | 54 (55) | 245 (252) | 75 (76)
Sciatica, parasthesia, blurred vision (Nervous system disorders) | 3 (3) | 0 (0) | 13 (13) | 2 (2) | 16 (16) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 3 (3)
Cough / Asthma (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 3 (3) | 37 (38) | 8 (8) | 52 (53) | 11 (11) — Asthma x 3, each in a different tx arm
Menstrual bleeding - heavy, inter, menometorrhagia (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 10 (10) | 2 (2) | 13 (13) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 5 (5) | 0 (0)
Nasopharyngitis / oropharangeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 12 (12) | 5 (5) | 13 (13) | 5 (5)
Rhinitis, rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 0 (0)
Pruritis / rash pruritic/ rash/ urticaria (Skin and subcutaneous tissue disorders) | 92 (92) | 22 (22) | 360 (367) | 67 (70) | 452 (459) | 89 (92)
Other skin conditions >0.1% (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 4 (4) | 1 (1) — Furuncle (2), hyperhidrosis (3)
Hypertension (Vascular disorders) | 22 (22) | 6 (6) | 1 (1) | 2 (2) | 23 (23) | 8 (8)
Hypotension (Vascular disorders) | 13 (13) | 5 (5) | 0 (0) | 1 (1) | 13 (13) | 6 (6)
Other vascular disorders > 0.1% (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 1 (1) — Hyperemia (3 - MOX+ALB) Rectal hemorrhage (1 - IVM +ALB)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor requires that the study results be published in their entirety prior to a PI presenting, publishing or otherwise communicating study results for an individual site

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT04311671/Prot_SAP_006.pdf